CLINICAL TRIAL: NCT04126980
Title: Early Discharged Lumbar Spine Fusion Reduced Postoperative Readmissions: A Follow-up Study in a National Cohort
Status: Completed | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2018-09-0006CC
Record Dates: First submitted 2019-09-22; First posted 2019-10-15 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Lumbar Spinal Fusion; Early Discharge; Readmission
MeSH Terms: interventions — Reoperation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ED group: The ED group who had less than 72 hours of hospitalization (including the preparation period which commonly took approximately 1 day) for the surgery.
  Interventions: Behavioral: Rates of readmission and reoperation
- Comparison group: The comparison group who were hospitalized for more than 72 hours but less than 12 days.
  Interventions: Behavioral: Rates of readmission and reoperation

INTERVENTIONS:
Behavioral: Rates of readmission and reoperation — All patients were then followed-up for 180 days after the indexed surgery of lumbar fusion. All-causes of re-hospitalization and re-operations for lumbar spine fusion, were analyzed at 30, 60 and 180 days for comparison between the ED group and the comparison group.

SUMMARY:
This study undertake to determine the effects of ED on readmissions and reoperations in lumbar fusion. The study enrolled patients who underwent lumbar fusion surgery at age 50-70 years from a national database, and grouped them into an ED group or a comparison group. All patients were then followed-up for 180 days after the indexed surgery of lumbar fusion.

DETAILED DESCRIPTION:
Surgery for lumbar fusion is one of the most commonly performed spinal arthrodesis procedures worldwide. In recent years, there has been the emerging popularity of strategies aimed at early discharge (ED) in such a field of spinal surgery. However, more data are required to corroborate the adaptation of ED in spinal surgery. The benefits of ED in lumbar fusion have not yet been validated by large cohort studies. This study undertake to determine the effects of ED on readmissions and reoperations in lumbar fusion.

This population-based retrospective cohort study used admission records of Taiwan's National Health Insurance Research Database (NHIRD). The NHIRD comprehensively contains de-identified claim data of Taiwan's National Health Insurance (NHI) program which covers 99% of the Taiwanese population and contracts with 97% of the providers of healthcare services in Taiwan. In order to protect privacy, the National Health Research Institute (NHRI) re-compiled, validated and de-identified the medical claims and finally made the data publicly available for medical researchers in Taiwan. In the admission database, the investigators are able to trace comprehensive information on the insured subjects, including gender, date of birth, dates of clinical visits and hospitalization, the International Classification of Diseases (Ninth Revision) Clinical Modification (ICD-9-CM) codes of diagnoses, ICD codes of surgical procedures, etc.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent lumbar spinal fusion surgery between July 2011 and June 2013 were identified and extracted in the NHIRD.

Exclusion Criteria:

* Inconsistent conditions

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent lumbar spinal fusion surgery between July 2011 and June 2013 were identified and extracted in the NHIRD.
Sampling Method: Non-Probability Sample
Enrollment: 18008 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2019-09-03 (Actual)

PRIMARY OUTCOMES:
Demographic characteristics | 2011-2013
  The comparison group and the ED group had some differences in gender composition, age, and medical comorbidities.

CONTACTS AND LOCATIONS:
Overall Officials: Taipei Veterans General Hospital, Study Director — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei County, Taiwan